CLINICAL TRIAL: NCT00301392
Title: Japan Prevention Trial of Diabetes by Pitavastatin in Patients With Impaired Glucose Tolerance (J-PREDICT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tokyo University (Other)
Responsible Party: Principal Investigator, Tsutomu Yamazaki, Professor, Tokyo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: J-PREDICT
Record Dates: First submitted 2006-03-05; First posted 2006-03-10 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Diabetes Mellitus; Glucose Intolerance
Keywords: Glucose intolerance; Diabetes mellitus; Statins,HMG-CoA
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pitavastatin (Other): Administration of Pitavastatin
  Interventions: Other: life-style intervention; Drug: Life style interventions plus concomitant use of pitavastatin.

INTERVENTIONS:
Other: life-style intervention — As the life-style interventions aiming to reduce the major risks of developing diabetes mellitus, instruct the following four items:(1)set diet right, (2)maintain normal weight,(3)improve physical activity,(4)normalize smoking and alcohol drinking.
Drug: Life style interventions plus concomitant use of pitavastatin. — Once-daily dosing of pitavastatin 1 mg(1 tablet of Livalo Tab 1 mg), or 2mg(2 tablets of Livalo Tab 1mg or 1 tablet of Livalo Tab 2mg);Dosing period of pitavastatin should be 60 months.(max.84 months).

SUMMARY:
The purpose of this study is to evaluate the effects of pitavastatin for preventing diabetes in a population with impaired glucose tolerance.

DETAILED DESCRIPTION:
Diabetes mellitus and its complications are major health problems globally. People with impaired glucose tolerance (IGT) are at high risk of developing diabetes. It is therefore important to focus on preventing diabetes in individuals with IGT. HMG-CoA reductase inhibitors (statins) are widely used for hypercholesterolemia, one of the most frequent metabolic disorders. However, there is no direct evidence to whether statins are beneficial for preventing diabetes. This study is designed to compare the efficacy of life-style modification versus life-style modification with pitavastatin (a statin) administration, in individuals with IGT.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for the screening test (within 6 months before screening):

* LDL-cholesterol 100-159 mg/dl and/or total cholesterol 180-239 mg/dl
* At least one of the following:

  1. Fasting plasma glucose 100-125 mg/dl, and/or casual (non-fasting) plasma glucose 120-199 mg/dl, and/or HbA1c 5.5-6.0%
  2. At least two of the following risk factors for impaired glucose tolerance:

     1. Second degree relative with diabetes
     2. BMI >= 24 kg/m2
     3. Systolic blood pressure >=130 mmHg, and/or diastolic blood pressure >= 85 mmHg, and/or receiving treatment for hypertension
     4. Triglyceride >= 150 mg/dl, and/or HDL < 40 mg/dl
* Written consent for participation in the study by their own volition after being provided sufficient explanation for the participation into this clinical trial

Inclusion Criteria for the entry (Confirmed by screening test):

-Impaired glucose tolerance by 75g oral glucose tolerance test (fasting plasma glucose <126 mg/dl and 2-h plasma glucose 140-199 mg/dl)

Exclusion Criteria:

* History of diabetes (except gestational diabetes)
* Fasting plasma glucose >= 126 mg/dl , and/or 2-h plasma glucose >= 200 mg/dl
* HbA1c >= 6.5%
* Diabetic retinopathy
* Receiving with hormone replacement therapy
* Pancreatic diseases ( e.g. pancreatitis, pancreatectomy, pancreatic cancer), Endocrine diseases ( e.g. Cushing's syndrome, acromegaly, pheochromocytoma, aldosteronism, hyperthyroidism )
* Receiving statins, fibrates or anion exchange resins
* Cancer or suspected cancer
* History of gastrectomy
* History of myocardial infarction, angina, or heart failure (NYHA Class >= III)
* Severe hypertension (SBP >= 180 mmHg or DBP >= 110 mmHg)
* Renal disease, including serum creatinine >= 2.0 mg/dl
* Hepatic disease, including transaminase (ALT or AST) >= 2 times the upper limit of normal
* Women hoping to become pregnant during the intended study period
* Contraindication or relative contraindication of Livalo® Tab(pitavastatin calcium)

  1. History of hypersensitivity to any of the ingredients of the product
  2. Severe hepatic disorder or biliary atresia
  3. Receiving cyclosporine
  4. Pregnant women, women suspected of being pregnant, or lactating women
  5. Patients receiving fibrates who also have laboratory evidence of abnormal renal function
* Familial hypercholesterolemia
* Drug abuse, alcoholism
* Individuals who are ineligible in the opinion of the investigator

Ages: 30 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1240 (Actual)
Dates: Start 2006-04; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of diabetes based on 1 positive OGTT or fasting glucose levels | from April, 2006 to end of March, 2012

SECONDARY OUTCOMES:
Incidence of newly developed diabetes | from April, 2006 to end of March, 2012
Cumulative incidence of diabetes based on clinical diagnosis. | from April, 2006 to end of March, 2012
  Cumulative incidence of diabetes based on clinical diagnosis defined as at least one of the following:(1) Typical symptoms of diabet plus 1 positive OGTT or fasting glucose levels, (2)HbA1c>=6.5% plus 1 positive OGTT or fasting glucose levels, (3)2 positive OGTT or fasting glucose levels.
Cumulative incidence of newly developed diabetes based on 1 positive OGTT or fasting glucose levels | from April, 2006 to end of March, 2012
  Cumulative incidence of newly developed diabetes based on 1 positive OGTT or fasting glucose levels (from the first administration of the study drug after the randomization)
Time until development of diabetes; Improvement in glucose tolerance | from April, 2006 to end of March, 2012
Incidence of any cardiovascular disease (myocardial infarction, angina, congestive heart disease, coronary revascularization, cerebral hemorrhage, cerebral infarction. | from April, 2006 to end of March, 2012
Incidence of coronary heart disease (myocardial infarction, angina, coronary revascularization) | from April, 2006 to end of March, 2012
Incidence of coronary heart disease plus cerebral infarction | from April, 2006 to end of March, 2012
LDL-cholesterol | from April, 2006 to end of March, 2012
HDL-cholesterol | from April, 2006 to end of March, 2012
Triglyceride | from April, 2006 to end of March, 2012
RLP-cholesterol | from April, 2006 to end of March, 2012
Adiponectin | from April, 2006 to end of March, 2012
High sensitive CRP | from April, 2006 to end of March, 2012
Asymmetrical dimethyl arginine (ADMA) | from April, 2006 to end of March, 2012
Urinary 8-OHd | from April, 2006 to end of March, 2012
Fasting plasma glucose | from April, 2006 to end of March, 2012
2-h plasma glucose during 75g oral glucose tolerance test | from April, 2006 to end of March, 2012
HbA1c | from April, 2006 to end of March, 2012
Insulin | from April, 2006 to end of March, 2012
HOMA-R | from April, 2006 to end of March, 2012
HOMA-β | from April, 2006 to end of March, 2012
Insulinogenic index | from April, 2006 to end of March, 2012
Time until dropout | from April, 2006 to end of March, 2012
Number of adverse events | from April, 2006 to end of March, 2012

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Kadowaki, MD,PhD, Study Chair — Professor, Department of Metabolic Diseases, Graduate School of Medicine, the University of Tokyo.
Locations (1):
- The University of Tokyo, Graduate School of Medicine, Bunkyo-ku, Tokyo, Japan